CLINICAL TRIAL: NCT03861234
Title: Safety, Tolerability and Pharmacodynamics of Single Rising Intravitreal and Multiple Rising Intravitreal Doses of BI 836880 in Patients With wAMD (Open Label, Non-randomized, Uncontrolled).
Brief Title: A Study to Test Different Doses of BI 836880 in Patients With an Eye Disease Called Wet Age-related Macular Degeneration (wAMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1336-0007; 2017-001221-40 (EudraCT Number)
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Wet Macular Degeneration
MeSH Terms: conditions — Wet Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 0.06 mg BI 836880 - SRD part (Experimental)
  Interventions: Drug: BI 836880
- 0.18 mg BI 836880 - SRD part (Experimental)
  Interventions: Drug: BI 836880
- 0.5 mg BI 836880 - SRD part (Experimental)
  Interventions: Drug: BI 836880
- 1 mg BI 836880 - SRD part (Experimental)
  Interventions: Drug: BI 836880
- 2 mg BI 836880 - SRD part (Experimental)
  Interventions: Drug: BI 836880
- 1 mg BI 836880 - cohort 1 MRD part (Experimental)
  Interventions: Drug: BI 836880
- 2 mg BI 836680 - cohort 2 MRD part (Experimental)
  Interventions: Drug: BI 836880
- 2 mg BI 836680 - cohort 3 MRD part (Experimental)
  Interventions: Drug: BI 836880

INTERVENTIONS:
Drug: BI 836880 — Solution for Intravitreal (IVT) injection

SUMMARY:
This is a study in people with an eye disease called wet age-related macular degeneration (wAMD). The purpose of the study is to find out how well different doses of a medicine called BI 836880 are tolerated.

People can participate if they are at least 55 years old and if they have new blood vessels in their eyes despite treatment (anti-VEGF therapies). The study has 2 parts. In the first part, people get only 1 dose of BI 836880. This part takes 6 weeks. In the second part, people get 3 times the same dose of BI 836880. This part takes 6 months. BI 836880 is injected into the eye. During the entire study doctors regularly check the health of the participants.

ELIGIBILITY:
Inclusion Criteria:

SRD part and MRD cohort 1 (treatment-resistant patients with wAMD):

* Men and women over the age of 55 with active Choroidal Neovascularisation (CNV) secondary to age-related macular degeneration (AMD) despite anti-Vascualr endothelial growth factor (VEGF) therapies (at least 3 prior injections with the last injection within 16 to 4 weeks before treatment). Active CNV secondary to AMD is to be defined either by recent fluorescein or optical coherence tomography (OCT) angiogram within 4 weeks prior to screening or fluorescein or OCT angiogram obtained prior to first anti VEGF-treatment to confirm the diagnosis and still active according to investigator judgement.
* For MRD part only: Central subfield retinal thickness >300 microns in the study eye on Heidelberg Spectralis Spectral Domain Optical Coherence Tomography (SD-OCT).
* Presence of sub- and/or intraretinal fluid on SD-OCT in the study eye.
* Any active CNV with subfoveal leakage in the study eye as determined by OCT
* No subretinal hemorrhage involving the fovea in the study eye.
* No significant subfoveal fibrosis or atrophy on SD-OCT in the study eye that, in the opinion of the investigator, is able to prevent improvement in best corrected visual acuity (BCVA) and/or central subfield thickness (CSFT).
* Best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) VA in the study eye between 75 and 24 letters inclusive (approximately 20/32 and 20/320 or 6/9.5 and 6/95) at screening.
* Best-corrected VA in the non-study eye better than best-corrected VA in the study-eye. If both eyes are eligible and have identical VA the investigator may select the study eye.
* Male or female patients. Women of childbearing potential (WOCBP) cannot be included. Men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.
* Signed informed consent consistent with ICH GCP guidelines and local legislation prior to participation in the trial, which includes medication washout and restrictions.
* Not under any administrative or legal supervision or under institutionalization due to regulatory or juridical order.

MRD cohort 2 (treatment-naive patients with wAMD):

* No subretinal hemorrhage involving the fovea in the study eye.
* No significant subfoveal fibrosis or atrophy on SD-OCT in the study eye that, in the opinion of the investigator, is able to prevent improvement in BCVA and/or CSFT.
* Male or female patients. Women of childbearing potential (WOCBP) cannot be included. Men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.
* Signed informed consent consistent with ICH GCP guidelines and local legislation prior to participation in the trial, which includes medication washout and restrictions.
* Not under any administrative or legal supervision or under institutionalization due to regulatory or juridical order.
* Men and women over the age of 55 with treatment-naïve CNV secondary to AMD.
* Any CNV with subfoveal activity in the study eye defined as evidence of sub- and/or intraretinal fluid, or subretinal hyper-reflective material, or angiographic leakage.
* Best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) VA in the study eye between 80 and 24 letters inclusive (approximately 20/25 and 20/320 or 6/7.5 and 6/95) at screening.
* Best-corrected ETDRS VA in the non-study eye 50 letters inclusive (approximately 20/100 or 6/30) or better at screening.
* If both eyes are eligible at screening, the study eye is the eye with the worse bestcorrected VA.

MRD cohort 3 (frequently treated patients):

* No subretinal hemorrhage involving the fovea in the study eye.
* No significant subfoveal fibrosis or atrophy on SD-OCT in the study eye that, in the opinion of the investigator and with the endorsement of the Sponsor, is able to prevent improvement in BCVA.
* Male or female patients. Women of childbearing potential (WOCBP)1 cannot be included.Men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.
* Signed informed consent consistent with ICH GCP guidelines and local legislation prior to participation in the trial, which includes medication washout and restrictions.
* Not under any administrative or legal supervision or under institutionalization due to regulatory or juridical order.
* Any CNV with subfoveal activity in the study eye defined as evidence of sub- and/or intraretinal fluid, or subretinal hyper-reflective material, or angiographic leakage.
* Best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) VA in the study eye between 80 and 24 letters inclusive (approximately 20/25 and 20/320 or 6/7.5 and 6/95) at screening.
* If both eyes are eligible at screening, the study eye is the eye with the worse bestcorrected VA.
* Men and women over the age of 55 with diagnosed wAMD that:

  * require frequent wAMD SoC (28-56 days between the last 3 treatments)
  * have had ≥ 3 previous treatments with IVT SoC (ranibizumab, aflibercept, or bevacizumab) in the study eye
  * had the last SoC injection ≥ 4 weeks, but no more than 8 weeks, before the first administration of the study drug
  * have been on SoC treatment ≥ 6 months and are within 3 years from initial wAMD diagnosis in the study eye

Exclusion criteria:

* Additional eye disease in the study eye that could compromise best corrected VA (BCVA) with visual field loss, uncontrolled glaucoma (intraocular pressure (IOP)> 24 mmHg on more than 2 consecutive measurements prior to screening), clinically significant diabetic maculopathy, history of ischemic optic neuropathy or retinalvascular occlusion, symptomatic vitreomacular traction, or genetic disorders such as retinitis pigmentosa); history of high myopia > 8 diopters in the study eye. Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation with SD-OCT.
* Any prior intraocular surgery in the study eye other then uneventful lens replacement for cataract within 3 months prior to screening.
* Aphakia or total absence of the posterior capsule. Yttrium aluminum garnet (YAG) laser capsulotomy permitted, more than 1 month prior to enrollment in the study eye.
* Current or planned use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoximine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol).
* Medical history or condition: Uncontrolled diabetes mellitus, with hemoglobin A1c (HbA1c) > 10%, myocardial infarction or stroke within 12 months of screening, active bleeding disorder, concomitant use of warfarin or anticoagulation therapy (use of antiplatelet therapy such as aspirin is allowed), major surgery within 1 month of screening or when planned within the study period, hepatic impairment, uncontrolled hypertension.
* Patients with a clinically relevant abnormal screening haematology, blood chemistry, or urinalysis, if the abnormality defines a significant disease as defined in other exclusion criteria. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 2.0-fold the upper limit of normal at screening. Patients with total bilirubin 2.5x upper limit of normal at screening.
* Patient with impaired renal function defined as calculated glomerular filtration rate (GFR) < 30 mL/min.
* Significant alcohol or drug abuse within past 2 years per investigator judgement.
* Further exclusion criteria apply.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (7):
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Verum Research, LLC, Eugene, Oregon
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Universitätsklinikum Ulm, Ulm
- United Kingdom (4):
  - Bristol Eye Hospital, Bristol
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital, London
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A non-randomised, uncontrolled, open label trial consisting of a single rising dose (SRD) part followed by a multiple rising dose (MRD) part. The SRD part and MRD cohort 1 included patients with treatment-resistant wet age-related macular degeneration (wAMD). Patients with treatment-naïve wAMD were included in MRD cohort 2 and patients within 3 years of initial wAMD were included in MRD cohort 3.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 0.06 mg BI 836880 - SRD Part: 0.06 mg BI 836880 solution for intravitreal (IVT) injection with diluent for BI 836880 concentrate for solution for injection 80mg/mL, 10 mL vial was administered as single IVT injection on Day 1, in patients with treatment-resistant wet age-related macular degeneration (wAMD).
- 0.18 mg BI 836880 - SRD Part: 0.18 mg BI 836880 solution for intravitreal (IVT) injection with diluent for BI 836880 concentrate for solution for injection 80mg/mL, 10 mL vial was administered as single IVT injection on Day 1, in patients with treatment-resistant wet age-related macular degeneration (wAMD).
- 0.5 mg BI 836880 - SRD Part: 0.5 mg BI 836880 solution for intravitreal (IVT) injection with diluent for BI 836880 concentrate for solution for injection 80mg/mL, 10 mL vial was administered as single IVT injection on Day 1, in patients with treatment-resistant wet age-related macular degeneration (wAMD).
- 1 mg BI 836880 - SRD Part: 1 mg BI 836880 solution for intravitreal (IVT) injection with diluent for BI 836880 concentrate for solution for injection 80mg/mL, 10 mL vial was administered as single IVT injection on Day 1, in patients with treatment-resistant wet age-related macular degeneration (wAMD).
- 2 mg BI 836880 - SRD Part: 2 mg BI 836880 solution for intravitreal (IVT) injection with diluent for BI 836880 concentrate for solution for injection 80mg/mL, 10 mL vial was administered as single IVT injection on Day 1, in patients with treatment-resistant wet age-related macular degeneration (wAMD).
- 1 mg BI 836880 - Cohort 1 MRD Part: 1 mg BI 836880 solution for intravitreal (IVT) injection with diluent for BI 836880 concentrate for solution for injection 80mg/mL, 10 mL vial was administered as three IVT injections on Day 1, Day 29 and Day 57, in patients with treatment-resistant wet age-related macular degeneration (wAMD).
- 2 mg BI 836680 - Cohort 2 MRD Part: 2 mg BI 836880 solution for intravitreal (IVT) injection with diluent for BI 836880 concentrate for solution for injection 80mg/mL, 10 mL vial was administered as three IVT injections on Day 1, Day 29 and Day 57, in patients with treatment-naïve wAMD.
- 2 mg BI 836680 - Cohort 3 MRD Part: 2 mg BI 836880 solution for intravitreal (IVT) injection with diluent for BI 836880 concentrate for solution for injection 80mg/mL, 10 mL vial was administered as three IVT injections on Day 1, Day 29 and Day 57, in patients within 3 years of initial wAMD.
Period: Overall Study
Arm/Group | 0.06 mg BI 836880 - SRD Part | 0.18 mg BI 836880 - SRD Part | 0.5 mg BI 836880 - SRD Part | 1 mg BI 836880 - SRD Part | 2 mg BI 836880 - SRD Part | 1 mg BI 836880 - Cohort 1 MRD Part | 2 mg BI 836680 - Cohort 2 MRD Part | 2 mg BI 836680 - Cohort 3 MRD Part
Started | 3 | 3 | 3 | 3 | 3 | 11 | 4 | 13
Treated | 3 | 3 | 3 | 3 | 3 | 10 | 4 | 13
Completed (Completed trial mediation) | 3 | 3 | 3 | 3 | 3 | 8 | 1 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Not completed — Not treated | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study medication discontinued due to safety notification | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — As per sponsor decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — IMP on hold as per sponsor instructions | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All patients who were treated with at least one dose of BI 836880.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.06 mg BI 836880 - SRD Part | 0.18 mg BI 836880 - SRD Part | 0.5 mg BI 836880 - SRD Part | 1 mg BI 836880 - SRD Part | 2 mg BI 836880 - SRD Part | 1 mg BI 836880 - Cohort 1 MRD Part | 2 mg BI 836680 - Cohort 2 MRD Part | 2 mg BI 836680 - Cohort 3 MRD Part | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 4 | 13 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 81.7 (5.7) | 76.7 (4.2) | 75.3 (1.5) | 75.7 (1.5) | 70.7 (1.2) | 77.0 (4.8) | 69.3 (13.0) | 77.0 (6.3) | 75.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 0 | 1 | 4 | 2 | 6 | 17
  Male | 1 | 1 | 3 | 3 | 2 | 6 | 2 | 7 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 10 | 4 | 13 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 3 | 10 | 4 | 13 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: SRD-part: Number of Participants With Ocular Dose Limiting Events (DLEs)
Description: Single rising dose (SRD)-part: Number of participants with ocular dose limiting events (DLEs).
Time Frame: From drug administration until the end of trial (EOT) visit in the SRD part, up to 6 weeks.
Population: Treated Set: All patients who were treated with at least on dose of BI 836880. SRD-part.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.06 mg BI 836880 - SRD Part | 0.18 mg BI 836880 - SRD Part | 0.5 mg BI 836880 - SRD Part | 1 mg BI 836880 - SRD Part | 2 mg BI 836880 - SRD Part
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: SRD-part: Number of Participants With Drug Related Adverse Events (AEs)
Description: Single rising dose (SRD)-part: Number of participants with drug related adverse events (AEs).
Time Frame: From drug administration until the end of trial (EOT) visit in the SRD part, up to 6 weeks.
Population: Treated Set (TS): All patients who were treated with at least one dose of BI 836680. SRD-part.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.06 mg BI 836880 - SRD Part | 0.18 mg BI 836880 - SRD Part | 0.5 mg BI 836880 - SRD Part | 1 mg BI 836880 - SRD Part | 2 mg BI 836880 - SRD Part
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: SRD-part: Number of Participants With Any Ocular Adverse Events in the Study Eye
Description: Single rising dose (SRD)-part: Number of participants with any ocular adverse events in the study eye.
Time Frame: From drug administration until the end of trial (EOT) visit in the SRD part, up to 6 weeks.
Population: Treated Set (TS): All patients who were treated with at least one dose of BI 836880. SRD-part.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.06 mg BI 836880 - SRD Part | 0.18 mg BI 836880 - SRD Part | 0.5 mg BI 836880 - SRD Part | 1 mg BI 836880 - SRD Part | 2 mg BI 836880 - SRD Part
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants | 1 | 0 | 1 | 1 | 2

4. Primary Outcome: MRD-part: Number of Participants With Drug Related Adverse Events (AEs)
Description: Multiple rising dose (MRD)-part: Number of participants with drug related adverse events (AEs)
Time Frame: From first drug administration until the end of trial (EOT) visit in the MRD part, up to 24 weeks.
Population: Treated Set: All patients who were treated with at least on dose of BI 836880. MRD-part.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg BI 836880 - Cohort 1 MRD Part | 2 mg BI 836680 - Cohort 2 MRD Part | 2 mg BI 836680 - Cohort 3 MRD Part
Number analyzed (Participants) | 10 | 4 | 13
Participants | 2 | 1 | 3

5. Secondary Outcome: MRD-part: Percentage Change From Baseline in Central Subfield Thickness (CSFT) in the Study Eye at Week 12
Description: Multiple rising dose (MRD)-part: Central subfield thickness was measured using Spectral domain-optical coherence tomography (SD-OCT) with the assessment performed by a qualified person and only specified OCT equipment was used. Optical coherence tomography angiography (OCT-A), a non-invasive imaging technique providing high-resolution volumetric blood flow information without the use of dye was also performed by a qualified person, and only specified device(s) were used. OCT images were sent to an independent CRC for evaluation. A detailed manual for OCT image acquisition and data transmission was provided. CSFT was investigated after 3 doses of BI 836880 in the MRD part of the trial at Week 12.
Time Frame: At baseline and at week 12.
Population: Full Analysis Set (FAS): All patients who were treated with at least one dose of BI 836880 and have baseline and on-treatment CSFT measurements for the study eye in the time interval from drug administration to Week 12. MRD part.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 1 mg BI 836880 - Cohort 1 MRD Part | 2 mg BI 836680 - Cohort 2 MRD Part | 2 mg BI 836680 - Cohort 3 MRD Part
Number analyzed (Participants) | 10 | 4 | 12
Percentage change | -7.7554 (18.9936) | -26.5552 (12.1400) | -0.1372 (20.1706)

6. Secondary Outcome: MRD-part: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye at Week 12
Description: Multiple rising dose (MRD)-part): Visual acuity (VA) measured by 'early treatment diabetic retinopathy study' letter charts.
  BCVA was measured using the early treatment diabetic retinopathy study (ETDRS) VA chart starting at a test distance of 4 m. The BCVA score was the number of letters read correctly by the patient. The assessment was performed by a trained person under specified conditions regarding examination room and equipment.
Time Frame: At baseline and at Week 12.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | 1 mg BI 836880 - Cohort 1 MRD Part | 2 mg BI 836680 - Cohort 2 MRD Part | 2 mg BI 836680 - Cohort 3 MRD Part
Number analyzed (Participants) | 10 | 4 | 13
Letters | -1.2 (6.4) | 1.8 (2.5) | -4.7 (22.3)

7. Secondary Outcome: MRD-part: Time to Recurrence in the Study Eye From Last Administration at Each Visit
Description: Multiple rising dose (MRD)-part: Time to recurrence was assessed in the MRD part from last trial drug administration to occurrence of any of the following in the study eye, leading to the use of wet age-related macular degeneration (wAMD) rescue medication as decided by the investigator:
  * Increase in Central Subfield Thickness (CFST) ≥75 μm with a decrease in Best Corrected Visual Acuity (BCVA) of ≥ 5 letters compared to Visit 5, OR
  * Decrease in BCVA of >5 letters compared to baseline (Visit 2), due to worsening wAMD activity, OR
  * Decrease in BCVA of ≥10 letters compared to the best prior BCVA, due to worsening wAMD activity From above criteria, if Visit 5 BCVA/CSFT assessment data is missing, BCVA/CSFT values available earlier than Visit 5 will be used. The last trial drug administration is strictly referring to the third injection, if a patient doesn't complete three injections, the patient will not be evaluated for time to recurrence endpoint and will be censored.
Time Frame: From last drug administration at Week 8 until End of Trial, up to 16 weeks.
Population: Treated Set (TS): All patients who were treated with at least one dose of BI 836880. MRD-part.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 1 mg BI 836880 - Cohort 1 MRD Part | 2 mg BI 836680 - Cohort 2 MRD Part | 2 mg BI 836680 - Cohort 3 MRD Part
Number analyzed (Participants) | 10 | 4 | 13
Weeks | 8.0 [4.6 to 16.1] | NA [NA to NA] — Median and confidence interval could not be calculated, as there was no event ("recurrence"). | NA [8.1 to NA] — Median and upper confidence interval could not be calculated, as all patients either censored or had events before the probability of recurrence reached to 50%.

8. Secondary Outcome: MRD-part: Number of Participants With Any Ocular Adverse Events in the Study Eye
Description: Multiple rising dose (MRD)-part: Number of participants with any ocular adverse events in the study eye.
Time Frame: From first drug administration until the end of trial (EOT) visit in the MRD part, up to 24 weeks.
Population: Treated Set (TS): All patients who were treated with at least one dose of BI 836880. MRD-part.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 mg BI 836880 - Cohort 1 MRD Part | 2 mg BI 836680 - Cohort 2 MRD Part | 2 mg BI 836680 - Cohort 3 MRD Part
Number analyzed (Participants) | 10 | 4 | 13
Participants | 5 | 1 | 9

ADVERSE EVENTS:
Time Frame: SRD-part: From drug administration until the end of trial (EOT) visit in the SRD part, up to 6 weeks. MRD-part: From first drug administration until the end of trial (EOT) visit in the MRD part, up to 24 weeks. All-cause mortality: Up to 6 weeks for SRD-part, up to 24 weeks for MRD-part.
Description: Treated Set (TS): All patients who were treated with at least one dose of BI 836880.
Arm/Group | 0.06 mg BI 836880 - SRD Part | 0.18 mg BI 836880 - SRD Part | 0.5 mg BI 836880 - SRD Part | 1 mg BI 836880 - SRD Part | 2 mg BI 836880 - SRD Part | 1 mg BI 836880 - Cohort 1 MRD Part | 2 mg BI 836680 - Cohort 2 MRD Part | 2 mg BI 836680 - Cohort 3 MRD Part
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/10 | 0/4 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 0/3 | 0/3 | 2/10 | 0/4 | 4/13
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/3 | 1/3 | 2/3 | 8/10 | 2/4 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.06 mg BI 836880 - SRD Part (N=3) | 0.18 mg BI 836880 - SRD Part (N=3) | 0.5 mg BI 836880 - SRD Part (N=3) | 1 mg BI 836880 - SRD Part (N=3) | 2 mg BI 836880 - SRD Part (N=3) | 1 mg BI 836880 - Cohort 1 MRD Part (N=10) | 2 mg BI 836680 - Cohort 2 MRD Part (N=4) | 2 mg BI 836680 - Cohort 3 MRD Part (N=13)
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Retinal occlusive vasculitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Depressed fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.06 mg BI 836880 - SRD Part (N=3) | 0.18 mg BI 836880 - SRD Part (N=3) | 0.5 mg BI 836880 - SRD Part (N=3) | 1 mg BI 836880 - SRD Part (N=3) | 2 mg BI 836880 - SRD Part (N=3) | 1 mg BI 836880 - Cohort 1 MRD Part (N=10) | 2 mg BI 836680 - Cohort 2 MRD Part (N=4) | 2 mg BI 836680 - Cohort 3 MRD Part (N=13)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anterior chamber cell (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lenticular opacities (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subretinal fluid (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitreal cells (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vitreous opacities (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Chorioretinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood folate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oxygen saturation abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tear break up time decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Labile hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT03861234/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT03861234/SAP_001.pdf